CLINICAL TRIAL: NCT04411472
Title: A DB, Placebo-Controlled, Two-Arm Parallel-Group, Phase 3 RCT to Investigate the Efficacy and Safety of Recombinant Human Alkaline Phosphatase for Treatment of Patients With SA-AKI
Brief Title: (Revival) Study to Investigate the Efficacy and Safety of Alkaline Phosphatase in Patients With Sepsis-Associated AKI
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Data Monitoring Committee (DMC) concluded that the pre-specified futility threshold was met and that there was no safety concern.
Sponsor: AM-Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP-recAP-AKI-03-01
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Results first posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Acute Kidney Injury Due to Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- active (Experimental): recombinant human alkaline phosphatase 1.6mg/kg 3 daily 1 hour infusions
  Interventions: Biological: Recombinant human alkaline phosphatase
- placebo (Placebo Comparator): matching placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Recombinant human alkaline phosphatase — patients with SA-AKI are randomly assigned in a 1:1 ratio to either placebo or 1.6 mg/kg recAP.
  Other Names: ilofotase alfa
  Arms: active
Other: Placebo — Placebo
  Arms: placebo

SUMMARY:
Clinical phase 3 study to investigate the effect of recAP on 28 day mortality in patients admitted to the ICU with acute kidney injury that is caused by sepsis.

The study has three distinct SA-AKI trial populations:

1. The main trial population: Patients with a pre-AKI reference eGFR ≥45 mL/min/1.73 m2 and no proven or suspected SARS-CoV-2 at time of randomization.
2. A 'moderate' CKD population: Patients with a pre-AKI reference eGFR ≥25 and <45 mL/min/1.73 m2 and no proven or suspected SARS-CoV-2 at time of randomization.
3. A Corona Virus Disease 2019 (COVID-19) population: Patients with proven or suspected SARS-CoV-2 at time of randomization with or without 'moderate' CKD. For patients in this population, COVID-19 should be the main cause of SA-AKI.

In the main study population approximately 1400 patients will be enrolled and in the two cohorts with moderate CKD and COVID-19 each up to 100 patients.

There are two arms in the study, one with active treatment and one with an inactive compound (placebo). Treatment is by 1 hour intravenous infusion, for three days. Patients are followed up for 28 days to see if there is an improvement on mortality, and followed for 90 and 180 days for mortality and other outcomes e.g. long-term kidney function and quality of life.

DETAILED DESCRIPTION:
Sepsis is the leading cause of acute kidney injury (AKI) and a major cause of death. Patients with SA-AKI have a high mortality and morbidity and are at risk of developing chronic kidney disease. AP is a homodimeric endogenous enzyme present in many cells and organs, e.g., intestines, placenta, liver, bone, kidney, and granulocytes. It exerts detoxifying effects through dephosphorylation of endotoxins; pathogen associated molecular pattern molecules (PAMPS e.g., lipopolysaccharide) and damage-associated molecular pattern molecules (DAMPS e.g., adenosine tri- and di-phosphate). In animal models of sepsis and AKI, administration of AP attenuates the inflammatory response, improves renal function and/or reduces mortality.

AM-Pharma B.V. is developing AP as a novel, recombinant chimeric human AP medicinal product, called recAP, to be used as an intravenous infusion for the treatment of SA-AKI. In the Phase 2 trial STOP-AKI, a survival benefit was observed in the two highest dose groups, 0.8 mg/kg and 1.6 mg/kg groups, compared to the placebo group. There were no safety or tolerability concerns for any of the doses tested (0.4, 0.8 and 1.6 mg/kg). The 1.6 mg/kg recAP dose was selected for this Phase 3 trial based on the significant survival benefit observed. PK/PD simulations also confirmed this dose to have the most pronounced treatment effect.

The primary objective of this Phase 3 trial is to confirm the mortality benefit seen in STOP-AKI by demonstrating a reduction in 28 day all cause mortality in patients with SA-AKI treated with 1.6 mg/kg recAP.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older.
2. In the ICU or intermediate care unit for clinical reasons.
3. Have sepsis requiring vasopressor (norepinephrine, epinephrine, dopamine, phenylephrine, vasopressin, or angiotensin II) therapy, i.e.:

   1. suspected or proven bacterial or viral infection. and
   2. on vasopressor therapy (≥0.1 µg/kg/min norepinephrine or equivalent) for sepsis-induced hypotension for at least one hour despite adequate fluid resuscitation according to clinical judgement. Following the initial one hour on at least 0.1 µg/kg/min norepinephrine or equivalent, any dose of vasopressor counts as vasopressor therapy.

   The combination of a) and b) automatically ensures that patients fulfill the Sepsis 3 criteria as 0.1 µg/kg/min norepinephrine corresponds to a score of +4 on the Cardiovascular sub-score of the SOFA score.
4. Have AKI according to at least one of the below KDIGO criteria, a to d:

   1. An absolute increase in serum or plasma creatinine (CR) by ≥0.3 mg/dL (≥26.5 µmol/L) within 48 hours.

      or
   2. A relative increase in CR to ≥1.5 times the pre-AKI reference CR value which is known or presumed to have occurred within prior 7 days.

      or
   3. A decrease in urinary output to <0.5 mL/kg/hour for a minimum of 6 hours following adequate fluid resuscitation.

   or d) If the patient does not have a known history of CKD and there is no pre-AKI reference CR value available from the past 12 months available from the past 12 months: a CR value greater or equal to the levels presented in Table 1, with the increase in CR presumed to have occurred within prior 7 days.
5. Provision of signed and dated ICF in accordance with local regulations.

Exclusion Criteria:

1. a) At sites where enrolment of 'moderate' CKD patients is allowed, patients with 'severe' CKD defined as a pre-AKI reference eGFR <25 mL/min/1.73 m2 are excluded.

   * For patients with known CKD, the most recent eGFR prior to index hospitalization needs to be documented as ≥25 mL/min/1.73 m2.
   * For patients with known CKD but no known eGFR prior to hospitalization, presentation eGFR between 25-60 mL/min/1.73 m2 can also be used to rule out 'severe' CKD.

     b) At sites where enrolment of 'moderate' CKD patients is NOT allowed, patients with 'moderate' and 'severe' CKD defined as a pre-AKI reference eGFR <45 mL/min/1.73 m2 are excluded.
   * For patients with known CKD, the most recent eGFR prior to index hospitalization needs to be documented as ≥45 mL/min/1.73 m2.
   * For patients with known CKD but no known eGFR prior to hospitalization, presentation eGFR between 45-60 mL/min/1.73 m2 can also be used to rule out 'moderate' and 'severe' CKD.
2. Advanced chronic liver disease, defined as a Child-Pugh score of 10 to 15 (Class C).
3. Acute pancreatitis without proven infection.
4. Urosepsis related to suspected or proven urinary tract obstruction.
5. Main cause of AKI not sepsis.
6. Proven or suspected SARS-CoV-2 infection. NOTE: This exclusion criterion does not apply to patients in the COVID-19 population, in which COVID-19 should be the main cause of SA-AKI.
7. Severe burns requiring ICU treatment.
8. Severely immunosuppressed, e.g. due to:

   * hematopoietic cell transplantation within past 6 months prior to Screening or acute or chronic graft-versus-host disease
   * solid organ transplantation
   * leukopenia not related to sepsis, i.e., preceding sepsis
   * Human Immunodeficiency Virus (HIV)/Acquired Immune Deficiency Syndrome (AIDS)
   * receiving chemotherapy within 30 days prior to Screening.
9. At high risk of being LTFU, e.g., due to known current or recent (within the last 6 months) IV drug abuse or known to be homeless.
10. Limitations to use of mechanical ventilation (MV), RRT or vasopressors and inotropes (NOTE: limitation of cardiopulmonary resuscitation (CPR) only is not an exclusion criterion).
11. Previous administration of recAP.
12. Use of a non-marketed drug within the last month or concurrent or planned participation in a clinical trial for a non-marketed drug or device. (NOTE: Co-enrollment or concurrent participation in observational, non-interventional trials using no protocolized treatments or procedures are always allowed. Co-enrollment or concurrent participation in trials using protocolized treatments or procedures, e.g. blood draws, requires pre-approval by the TSC).
13. Current or planned extracorporeal membrane oxygenation (ECMO).
14. On RRT >24 hours before start of trial drug.
15. No longer on vasopressor therapy at time of randomization.
16. On continuous vasopressor therapy for >72 hours before start of trial drug.
17. Estimated glomerular filtration rate (eGFR) >60 mL/min/1.73 m2 based on the most recent available CR sample at time of screening (NOTE: will often be the sample used to diagnose AKI). eGFR should be calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula. In Japan, the CKD-EPI formula with Japanese coefficient should be used. If local regulations prohibit correcting for race in the calculation of eGFR, it is acceptable to use the formula without correcting for race.
18. Not feasible to start trial drug within:

    1. 48 hours from AKI diagnosis, when AKI diagnosis precedes start of vasopressor therapy.

       or
    2. 24 hours from AKI diagnosis, when AKI is diagnosed after start of vasopressor therapy.
19. Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 676 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A Legters, Study Director — AM-Pharma
Locations (122):
- United States (16):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - The George Washington University Medical Faculty Associates - Anesthesiology, Washington D.C., District of Columbia
  - Emory Clinical Cardiovascular Research Institute, Atlanta, Georgia
  - Glenbrook Hospital, Glenview, Illinois
  - NorthShore Medical Group - Bannockburn, Highland Park, Illinois
  - University of Kentucky College of Medicine (UKCM), Lexington, Kentucky
  - Regions Hospital, Saint Paul, Minnesota
  - University of New Mexico School of Medicine, Albuquerque, New Mexico
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - The Ohio State University - Dorothy M. Davis Heart and Lung Research Institute, Columbus, Ohio
  - UPMC CancerCenter at Magee - Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - University of Virginia Health System, Charlottesville, Virginia
  - Froedtert & the Medical College of Wisconsin Froedtert Hospital, Milwaukee, Wisconsin
- Australia (7):
  - Flinders Medical Centre, Bedford Park
  - Bendigo Hospital, Bendigo
  - Footscray Hospital, Footscray
  - Austin Hospital, Melbourne
  - John Hunter Hospital, New Lambton Heights
  - Sunshine Hospital ICU - Western Hospital, Saint Albans
  - Gold Coast University Hospital (GCUH), Southport
- Austria (3):
  - Medizinische Universitaet Graz - Klinik fuer Innere Medizin, Graz
  - Medizinische Universitaet Innsbruck - Universitaetsklinik fuer Innere Medizin I, Innsbruck
  - Medizinische Universität Innsbruck, Innsbruck
- Belgium (9):
  - Centre Hospitalier Universitaire Brugmann, Brussels
  - Centre Hospitalier Universitaire (CHU) de Charleroi - Hopital Civil Marie Curie, Charleroi
  - Ziekenhuis Oost-Limburg, Genk
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Brussel, Jette
  - Hôpital de JOLIMONT, La Louvière
  - Clinique Saint-Pierre- Ottignies, Ottignies
  - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert
  - CHU UCL Namur - Mont-Godinne, Yvoir
- Canada (10):
  - Peter Lougheed Centre, Calgary
  - Foothills Medical Centre, Calgary
  - Rockyview General Hospital, Calgary
  - Alberta Health Services - South Health Campus Hospital, Calgary
  - The Ottawa Hospital - General Campus, Ottawa
  - The Ottawa Hospital - Civic Campus, Ottawa
  - Hôpital de l'Enfant-Jésus, Québec
  - St. Paul's Hospital, Vancouver
  - Royal Jubilee Hospital (RJH), Victoria
  - Victoria General Hospital (VGH), Victoria
- Denmark (10):
  - Aalborg Universitetshospital, Aalborg
  - Aarhus University Hospital, Aarhus N
  - Rigshospitalet, Copenhagen
  - Herning Regional Hospital, Herning
  - Nordsjællands Hospital, Hillerød
  - Sjaellands Universitetshospital, Koge - Kardiologisk Afdeling, Køge
  - Odense Universitetshospital, Odense C
  - Regionshospitalet Randers, Randers
  - Slagelse Sygehus, Slagelse
  - Hospitalsenhed Midt, Viborg
- Finland (3):
  - Helsinki University Central Hospital (HUCH), Helsinki
  - Tampere University Hospital, Tampere
  - Turku University Hospital (TYKS), Turku
- France (16):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Centre Hospitalier d'Argenteuil, Argenteuil
  - Centre Hospitalier de Bethune Germon et Gauthier, Béthune
  - Centre Hospitalier René-Dubos, Cergy-Pontoise
  - CHU Dijon - Hôpital François Mitterrand, Dijon
  - Centre Hospitalier Départemental de Vendée - Les Oudairies, La Roche-sur-Yon
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Centre Hospitalier du Mans, Le Mans
  - CHU Limoges - Hôpital Dupuytren, Limoges
  - CHU de Nancy, Nancy
  - CHU de Nantes - Hôtel-Dieu, Nantes
  - CHU de Nimes - Hopital Universitaire Caremeau, Nîmes
  - Hôpital La Source, Orléans
  - Hôpital Lariboisière, Paris
  - Hôpitaux Universitaires de Strasbourg - Hôpital Civil, Strasbourg
  - CHRU de Tours - Hôpital Bretonneau, Tours
- Germany (5):
  - Universitätsklinikum Aachen, Aachen
  - Universitätsklinikum Hamburg-Eppendorf (UKE), Hamburg
  - University Hospital Jena - Klinik fur Neurologie, Jena
  - Universitaetsklinikum Leipzig - Klinik und Poliklinik fuer Gastroenterologie und Rheumatologie, Leipzig
  - University Hospital Münster, Münster
- Ireland (4):
  - National University of Ireland, Galway, Galway, G
  - St. James's Hospital, Dublin
  - Tallaght University Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
- Japan (11):
  - Tokyo Medical University Hachioji Medical Center, Hachioji-Shi
  - Hiroshima University Hospital, Hiroshima
  - Aso Iizuka Hospital, Izuka-shi
  - Rinku General Medical Center, Izumisano
  - Nara Medical University Hospital, Kashihara-shi
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Osaka City General Hospital, Osaka
  - Osaka Police Hospital, Osaka
  - Omihachiman Community Medical Center, Ōmihachiman
  - Fujita Health University Hospital, Toyoake-Shi
  - National Hospital Organization - Yokohama Medical Center, Yokohama
- Netherlands (7):
  - Jeroen Bosch Ziekenhuis lokatie GZG, 's-Hertogenbosch, North Brabant
  - Amsterdam UMC - VUMC, Amsterdam
  - Ziekenhuis Gelderse Vallei, Ede
  - Medisch Spectrum Twente, Enschede
  - Zuyderland Medisch Centrum, Heerlen, Heerlen
  - Radboud UMC, Nijmegen
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
- New Zealand (8):
  - Wellington Hospital, Wellington, WGN
  - Auckland City Hospital, Auckland
  - Middlemore Clinical Trials, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Auckland City Hospital, Grafton
  - Hawke's Bay Hospital Soldiers' Memorial, Hastings
  - Lakes District Health Board - Rotorua Hospital, Rotorua
- Spain (8):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitari de Bellvitge (IDIBELL), Barcelona
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital Clínico San Carlos, Madrid
  - Parc Taulí Sabadell Hospital Universitari, Sabadell
  - Universitat de Barcelona - Hospital Universitari Mutua Terrassa (HUMT), Terrassa
- United Kingdom (5):
  - University College London Hospitals NHS Foundation Trust - University College Hospital, London, LND
  - University Hospital of Wales, Cardiff
  - Royal Liverpool University Hospital, Liverpool
  - Guy's and St Thomas' NHS Foundation Trust - St Thomas' Hospital, London
  - Plymouth Hospitals NHS Trust - Derriford Hospital, Plymouth

REFERENCES:
- [Result] Pickkers P, Angus DC, Bass K, Bellomo R, van den Berg E, Bernholz J, Bestle MH, Doi K, Doig CJ, Ferrer R, Francois B, Gammelager H, Pedersen UG, Hoste E, Iversen S, Joannidis M, Kellum JA, Liu K, Meersch M, Mehta R, Millington S, Murray PT, Nichol A, Ostermann M, Pettila V, Solling C, Winkel M, Young PJ, Zarbock A; REVIVAL investigators. Phase-3 trial of recombinant human alkaline phosphatase for patients with sepsis-associated acute kidney injury (REVIVAL). Intensive Care Med. 2024 Jan;50(1):68-78. doi: 10.1007/s00134-023-07271-w. Epub 2024 Jan 3. PMID 38172296
- [Result] Pickkers P, Angus DC, Arend J, Bellomo R, van den Berg E, Bernholz J, Bestle M, Broglio K, Carlsen J, Doig CJ, Ferrer R, Joannidis M, Francois B, Doi K, Kellum JA, Laterre PF, Liu K, Mehta RL, Murray PT, Ostermann M, Pettila V, Richards S, Young P, Zarbock A, Kjolbye AL. Study protocol of a randomised, double-blind, placebo-controlled, two-arm parallel-group, multi-centre phase 3 pivotal trial to investigate the efficacy and safety of recombinant human alkaline phosphatase for treatment of patients with sepsis-associated acute kidney injury. BMJ Open. 2023 Apr 3;13(4):e065613. doi: 10.1136/bmjopen-2022-065613. PMID 37012016

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The target participant population consisted of adult participants in the intensive care unit or intermediate care unit with sepsis and new, recent onset acute kidney injury.
Pre-assignment Details: 676 participants were enrolled; 21 were screening failures and were not randomized. 5 participants (2 in the active group and 3 in the placebo group) were randomized, but not been exposed to any trial drug. Consequently, 650 patients have been randomized and treated (modified ITT population according to protocol). The mITT population is the basis for the primary efficacy analysis and most of the secondary analyses reported in clintrials.gov (1-6,8-16).
Groups:
- Placebo (Main Trial Population): Matching placebo; 3 daily 1-hour continuous intravenous infusions on Days 1, 2 and 3.
  Main Trial Population: Participants with a pre-AKI reference eGFR greater than or equal to 45 mL/min/1.73 m2 and no proven or suspected COVID-19 at time of randomization
- recAP 1.6 mg/kg (Main Trial Population): Recombinant human alkaline phosphatase (recAP) 1.6mg/kg; 3 daily 1-hour continuous intravenous infusions on Days 1, 2 and 3
  Main Trial Population: Participants with a pre-AKI reference eGFR greater than or equal to 45 mL/min/1.73 m2 and no proven or suspected COVID-19 at time of randomization
- Placebo (Moderate CKD Population): Matching placebo; 3 daily 1-hour continuous intravenous infusions on Days 1, 2 and 3.
  Moderate chronic kidney disease (CKD) Population: Participants with a pre-acute kidney injury reference estimated glomerular filtration rate more than or equal to 25 and less than 45 mL/min/1.73 m2 and no proven or suspected COVID-19 at time of randomization
- recAP 1.6 mg/kg (Moderate CKD Population): Recombinant human alkaline phosphatase (recAP) 1.6mg/kg; 3 daily 1-hour continuous intravenous infusions on Days 1, 2 and 3
  Moderate chronic kidney disease (CKD) Population: Participants with a pre-acute kidney injury reference estimated glomerular filtration rate more than or equal to 25 and less than 45 mL/min/1.73 m2 and no proven or suspected COVID-19 at time of randomization
- Placebo (COVID-19 Population): Matching placebo; 3 daily 1-hour continuous intravenous infusions on Days 1, 2 and 3.
  COVID-19 Population: Participants with proven or suspected COVID-19 at time of randomization with or without 'moderate' chronic kidney disease and, for patients in this population, COVID-19 should have been the main cause of sepsis-associated acute kidney injury
- recAP 1.6 mg/kg (COVID-19 Population): Recombinant human alkaline phosphatase (recAP) 1.6mg/kg; 3 daily 1-hour continuous intravenous infusions on Days 1, 2 and 3
  COVID-19 Population: Participants with proven or suspected COVID-19 at time of randomization with or without 'moderate' chronic kidney disease and, for patients in this population, COVID-19 should have been the main cause of sepsis-associated acute kidney injury
Period: Overall Study
Arm/Group | Placebo (Main Trial Population) | recAP 1.6 mg/kg (Main Trial Population) | Placebo (Moderate CKD Population) | recAP 1.6 mg/kg (Moderate CKD Population) | Placebo (COVID-19 Population) | recAP 1.6 mg/kg (COVID-19 Population)
Started | 277 | 279 | 31 | 30 | 13 | 20
Completed | 253 | 248 | 27 | 29 | 13 | 20
Not Completed | 24 | 31 | 4 | 1 | 0 | 0
Not completed — Adverse Event | 5 | 10 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 17 | 20 | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for the modified intent-to-treat population
Groups:
- Placebo (Main Trial Population): Matching placebo; 3 daily 1-hour continuous intravenous infusions on Days 1, 2 and 3
  Main Trial Population: Participants with a pre-AKI reference eGFR greater than or equal to 45 mL/min/1.73 m2 and no proven or suspected COVID-19 at time of randomization
- Total: Total of all reporting groups
Arm/Group | Placebo (Main Trial Population) | recAP 1.6 mg/kg (Main Trial Population) | Placebo (Moderate CKD Population) | recAP 1.6 mg/kg (Moderate CKD Population) | Placebo (COVID-19 Population) | recAP 1.6 mg/kg (COVID-19 Population) | Total
Number analyzed (Participants) | 277 | 279 | 31 | 30 | 13 | 20 | 650
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (12.73) | 68.4 (10.94) | 73.2 (8.90) | 70.2 (11.28) | 68.8 (7.67) | 62.8 (10.35) | 68.0 (11.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 105 | 8 | 12 | 2 | 6 | 237
  Male | 173 | 174 | 23 | 18 | 11 | 14 | 413
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 23 | 16 | 0 | 0 | 1 | 1 | 41
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 6 | 0 | 1 | 0 | 3 | 19
  White | 227 | 233 | 27 | 26 | 11 | 15 | 539
  More than one race | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 18 | 22 | 4 | 3 | 1 | 1 | 49
Height [Mean (Standard Deviation); unit: centimeters] — Population: The height and weight information was missing for one participant in the placebo group.
  centimeters
    number analyzed (Participants) | 276 | 279 | 31 | 30 | 13 | 20 | 649
    (all) | 170.4 (10.20) | 170.5 (10.30) | 171.2 (8.84) | 171.8 (8.98) | 170.0 (10.13) | 174.3 (10.06) | 170.7 (10.12)
Weight [Mean (Standard Deviation); unit: kilograms] — Population: The height and weight information was missing for one participant in the placebo group.
  kilograms
    number analyzed (Participants) | 276 | 279 | 31 | 30 | 13 | 20 | 649
    (all) | 86.9 (26.23) | 87.9 (25.67) | 87.3 (17.08) | 86.5 (16.94) | 98.9 (26.67) | 87.1 (19.39) | 87.6 (25.06)
Acute Physiology and Chronic Health Evaluation II total score [Mean (Standard Deviation); unit: score] — The Acute Physiology and Chronic Health Evaluation (APACHE) II score is a severity-of-disease classification system, used in ICU or intermediate care unit settings. A score from 0 to 71 was calculated in the eCRF from 12 physiological measurements using the worst value within the past 24 hours, age, and chronic health points (history of system organ failure). Higher scores indicate more severe disease and higher mortality risk. The score was calculated based on values from the 24 hours up to time of randomization Population: The score was not recorded for 25 participants. This included 10 participants in the placebo group (main trial population), 13 participants in the recAP 1.6 mg/kg group (main trial population), 1 participant in the recAP 1.6 mg/kg group (moderate CKD population), and 1 participant in the recAP 1.6 mg/kg group (COVID-19 population).
  score
    number analyzed (Participants) | 267 | 266 | 31 | 29 | 13 | 19 | 625
    (all) | 23.2 (7.17) | 23.2 (7.65) | 25.8 (7.00) | 23.6 (5.77) | 23.1 (6.87) | 23.6 (8.31) | 23.3 (7.34)
Modified sequential organ failure assessment total score (eCRF) [Mean (Standard Deviation); unit: score] — The Modified Sequential Organ Failure Assessment Score (mSOFA score) consists of 5 subscores (respiration, coagulation, Liver function, cardiovascular function and renal function) each ranging from 0=normal to 4=most abnormal. mSOFA is the sum of the 5 subscores (ranging from 0=normal in all subscores to 20=most abnormal in all subscores). The modified SOFA score used in the trial is exclusive of the 6th subscore (Central nervous system) from the original SOFA score published by Vincent at al. (1996). Population: The score was not recorded for 1 participant in the placebo group and 3 participants in the recAP 1.6 mg/kg group (main trial population).
  score
    number analyzed (Participants) | 276 | 276 | 31 | 30 | 13 | 20 | 646
    (all) | 9.4 (2.52) | 9.1 (2.33) | 9.5 (1.46) | 9.0 (1.88) | 9.4 (1.66) | 9.6 (2.03) | 9.3 (2.34)
Pre-acute kidney injury reference creatinine [Mean (Standard Deviation); unit: μmol/L] — Population: The value was not recorded for 1 participant in the placebo group.
  μmol/L
    number analyzed (Participants) | 276 | 279 | 31 | 30 | 13 | 20 | 649
    (all) | 83.36 (22.316) | 82.23 (21.865) | 130.42 (56.751) | 122.56 (33.684) | 87.99 (23.494) | 95.97 (27.159) | 87.42 (28.542)
Pre-acute kidney injury reference estimated glomerular filtration rate [Mean (Standard Deviation); unit: mL/min/1.73 m²] — Population: The value was not recorded for 1 participant in the placebo group.
  mL/min/1.73 m²
    number analyzed (Participants) | 276 | 279 | 31 | 30 | 13 | 20 | 649
    (all) | 76.16 (18.160) | 76.35 (18.059) | 52.36 (25.715) | 51.57 (21.945) | 74.88 (15.742) | 72.82 (18.438) | 73.84 (19.917)
Acute kidney injury diagnosis creatinine [Mean (Standard Deviation); unit: μmol/L] — Population: The diagnosis was not recorded for 1 participant in the placebo group.
  μmol/L
    number analyzed (Participants) | 276 | 279 | 31 | 30 | 13 | 20 | 649
    (all) | 212.43 (138.656) | 200.06 (123.685) | 270.10 (286.051) | 210.11 (93.540) | 176.20 (42.570) | 211.30 (148.803) | 209.00 (140.799)
Acute kidney injury diagnosis estimated glomerular filtration rate [Mean (Standard Deviation); unit: mL/min/1.73 m²] — Population: The diagnosis was not recorded for 1 participant in the placebo group.
  mL/min/1.73 m²
    number analyzed (Participants) | 276 | 279 | 31 | 30 | 13 | 20 | 649
    (all) | 32.28 (14.888) | 33.10 (14.958) | 25.93 (12.042) | 30.97 (20.116) | 33.54 (7.002) | 35.42 (16.461) | 32.39 (15.045)
KDIGO Chronic Kidney Disease stage [Count of Participants; unit: Participants] — KDIGO CKD staging:
  1. Normal or high (greater than or equal to 90 mL/min/1.73 min^2)
  2. Mildly decreased (greater than or equal to 60 and less than 90 mL/min/1.73m^2)
  3a: Mildly to moderately decreased (greater than or equal to 45 and less than 60 mL/min/1.73m^2)
  3b: Moderately to severely decreased (greater than or equal to 30 and less than 45 mL/min/1.73m^2)
  4: Severely decreased (greater than or equal to 15 and less than 30 mL/min/1.73m^2)
  5: Kidney failure (less than 15 mL/min/1.73m^2)
  From KDIGO 2012 Clinical Practice Guideline for the Evaluation and Management of CKD
  Participants
    1 | 67 | 69 | 4 | 2 | 3 | 3 | 148
    2 | 152 | 153 | 6 | 9 | 8 | 13 | 341
    3a | 53 | 50 | 2 | 0 | 2 | 3 | 110
    3b | 3 | 7 | 15 | 17 | 0 | 0 | 42
    4 | 1 | 0 | 3 | 2 | 0 | 1 | 7
    5 | 0 | 0 | 1 | 0 | 0 | 0 | 1
    Missing | 1 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: 28-day All-cause Mortality: Main Trial Population
Description: To demonstrate an effect of recAP on 28 day all cause mortality
Time Frame: 28 days
Population: Main Trial modified intent-to-treat Population
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Matching placebo; 3 daily 1-hour continuous intravenous infusions on Days 1, 2 and 3
- recAP 1.6 mg/kg: Recombinant human alkaline phosphatase (recAP) 1.6mg/kg; 3 daily 1-hour continuous intravenous infusions on Days 1, 2 and 3
Arm/Group | Placebo | recAP 1.6 mg/kg
Number analyzed (Participants) | 277 | 279
Participants
  Participants with known survival status at Day 28 | 272 | 279
  Number of participants died by Day 28 | 69 | 80
  Participants where survival status is unknown at Day 28 | 5 | 0
Statistical Analysis 1: Comparison: Placebo vs recAP 1.6 mg/kg; Test type: Superiority; p = 0.8025, One-sided p-value; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.805 to 1.732]

2. Primary Outcome: 28-day All-cause Mortality: Moderate Chronic Kidney Disease Population
Description: To demonstrate an effect of recAP on 28 day all cause mortality
Time Frame: 28 days
Population: Moderate Chronic Kidney Disease modified intent-to-treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | recAP 1.6 mg/kg
Number analyzed (Participants) | 31 | 30
Participants
  Participants with known survival status at Day 28 | 31 | 29
  Number of participants died by Day 28 | 10 | 6
  Participants where survival status is unknown at Day 28 | 0 | 1
Statistical Analysis 1: Comparison: Placebo vs recAP 1.6 mg/kg; Test type: Superiority; p = 0.1824, One-sided p-value; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.139 to 2.131]

3. Primary Outcome: 28-day All-cause Mortality: COVID-19 Population
Description: To demonstrate an effect of recAP on 28 day all cause mortality
Time Frame: 28 days
Population: COVID-19 modified intent-to-treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | recAP 1.6 mg/kg
Number analyzed (Participants) | 13 | 20
Participants
  Participants with known survival status at Day 28 | 13 | 20
  Number of participants died by Day 28 | 11 | 5
  Participants where survival status is unknown at Day 28 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs recAP 1.6 mg/kg; Test type: Superiority; p = 0.0080, One-sided p-value; Odds Ratio (OR) = 0.02, 95% CI 2-sided [0.001 to 0.405]

4. Secondary Outcome: Major Adverse Kidney Events 90: Main Trial Population
Description: Major adverse kidney events (MAKE) 90: dead by Day 90 or on Renal Replacement Therapy (RRT) at Day 90 or greater than or equal to 25% decline in estimated glomerular filtration rate (eGFR) on both Day 28 and Day 90 relative to the known or assumed pre-acute kidney injury reference level.
Time Frame: 90 Days
Population: Main Trial modified intent-to-treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | recAP 1.6 mg/kg
Number analyzed (Participants) | 277 | 279
Participants
  Participants with missing data on MAKE 90 | 36 | 49
  Participants with unknown data on MAKE 90 | 46 | 34
  MAKE 90: Dead | 89 | 97
  MAKE 90: On RRT | 2 | 0
  MAKE 90: greater than or equal to 25% decline in eGFR rate on both Day 28 and Day 90 | 15 | 7
Statistical Analysis 1: Comparison: Placebo vs recAP 1.6 mg/kg; Test type: Superiority; p = 0.3894, One-sided p-value; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.606 to 1.454]

5. Secondary Outcome: Major Adverse Kidney Events 90: Moderate Chronic Kidney Disease Population
Description: as for outcome 4
Time Frame: 90 Days
Population: Moderate Chronic Kidney Disease modified intent-to-treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | recAP 1.6 mg/kg
Number analyzed (Participants) | 31 | 30
Participants
  Participants with missing data on MAKE 90 | 7 | 7
  Participants with unknown data on MAKE 90 | 2 | 6
  MAKE 90: Dead | 13 | 7
  MAKE 90: On RRT | 0 | 0
  MAKE 90: greater than or equal to 25% decline in eGFR rate on both Day 28 and Day 90 | 1 | 1
Statistical Analysis 1: Comparison: Placebo vs recAP 1.6 mg/kg; Test type: Superiority; p = 0.1237, One-sided p-value; Odds Ratio (OR) = 0.47, 95% CI 2-sided [0.128 to 1.697]

6. Secondary Outcome: Major Adverse Kidney Events 90: COVID-19 Population
Description: as for outcome 4
Time Frame: 90 Days
Population: COVID-19 modified intent-to-treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | recAP 1.6 mg/kg
Number analyzed (Participants) | 13 | 20
Participants
  Participants with missing data on MAKE 90 | 1 | 4
  Participants with unknown data on MAKE 90 | 0 | 0
  MAKE 90: Dead | 11 | 6
  MAKE 90: On RRT | 0 | 0
  MAKE 90: greater than or equal to 25% decline in eGFR rate on both Day 28 and Day 90 | 1 | 0

7. Secondary Outcome: Major Adverse Kidney Events Through Day 90: Combined Population
Description: Major Adverse Kidney Events through day 90 (MAKE90A) :
  * death until day 90
  * greater than 25% drop in estimated glomerular filtration rate at Day 90
  * on renal replacement therapy (RRT) at day 90 OR on RRT through Day 28
Time Frame: 90 Days
Population: Combined population: From the 650 patients in the mITT population (321 Placebo and 329 recAP), 649 were analysed in the combined population (1 participant randomized and treated with placebo has been excluded as no efficacy data were available). In the combined population participants were analyzed as treated, resulting in 319 Placebo and 330 recAP participants (2 participants randomized to Placebo were treated with recAP, 1 participant randomized to recAP was treated with placebo).
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Matching placebo; 3 daily 1-hour continuous intravenous infusions on Days 1, 2 and 3 (Combined Population)
- recAP 1.6 mg/kg: Recombinant human alkaline phosphatase (recAP) 1.6mg/kg; 3 daily 1-hour continuous intravenous infusions on Days 1, 2 and 3 (Combined Population)
Arm/Group | Placebo | recAP 1.6 mg/kg
Number analyzed (Participants) | 319 | 330
Participants
  MAKE90A | 206 | 187
  Death until day 90 | 111 | 112
  Greater than 25% drop in eGFR at Day 90 visit | 28 | 19
  On RRT at Day 90 visit OR on RRT through day 28 | 116 | 93
  Rehospitalization | 30 | 28
Statistical Analysis 1: Comparison: Placebo vs recAP 1.6 mg/kg; Test type: Superiority; p = 0.019, one-sided p-value — one-sided p-value based on the z-score statistic for the difference in proportions; z-score statistic difference proportions = -7.9, 95% CI 2-sided [-15.4 to -0.4]

8. Secondary Outcome: Days Alive and Free of Organ Support Through Day 28: Main Trial Population
Description: Days alive and free of organ support through Day 28, ie, days alive with no mechanical ventilation (MV), Renal Replacement Therapy (RRT), vasopressors, or inotropes (with death within 28 days counting as zero days)
Time Frame: 28 days
Population: Main Trial modified intent-to-treat Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | recAP 1.6 mg/kg
Number analyzed (Participants) | 277 | 279
days
  Days alive and free of organ support through to Day 28 | 13.2 (11.33) | 12.8 (11.34)
  Number of days free of MV | 14.7 (11.93) | 14.3 (12.19)
  Number of days free of RRT | 18.4 (12.40) | 17.9 (12.64)
  Number of days free of vasopressors and inotropes | 16.5 (10.85) | 15.9 (11.17)
Statistical Analysis 1: Comparison: Placebo vs recAP 1.6 mg/kg; Days alive and free of organ support through to Day 28; Test type: Superiority; p = 0.5460, One-sided p-value from re-randomization
Statistical Analysis 2: Comparison: Placebo vs recAP 1.6 mg/kg; Number of days free of MV; Test type: Superiority; p = 0.6770, One-sided p-value from re-randomization
Statistical Analysis 3: Comparison: Placebo vs recAP 1.6 mg/kg; Number of days free of RRT; Test type: Superiority; p = 0.9930, One-sided p-value from re-randomization
Statistical Analysis 4: Comparison: Placebo vs recAP 1.6 mg/kg; Number of days free of vasopressors and inotropes; Test type: Superiority; p = 0.7790, One-sided p-value from re-randomization

9. Secondary Outcome: Days Alive and Free of Organ Support Through Day 28: Moderate Chronic Kidney Disease Population
Description: as for outcome 8
Time Frame: 28 days
Population: Moderate Chronic Kidney Disease modified intent-to-treat Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | recAP 1.6 mg/kg
Number analyzed (Participants) | 31 | 30
days
  Days alive and free of organ support through to Day 28 | 10.5 (10.59) | 17.2 (10.39)
  Number of days free of MV | 11.2 (11.47) | 18.1 (11.11)
  Number of days free of RRT | 17.8 (12.81) | 21.4 (11.71)
  Number of days free of vasopressors and inotropes | 14.8 (11.15) | 19.4 (10.58)
Statistical Analysis 1: Comparison: Placebo vs recAP 1.6 mg/kg; Days alive and free of organ support through Day 28; Test type: Superiority; p = 0.0510, One-sided p-value from re-randomization
Statistical Analysis 2: Comparison: Placebo vs recAP 1.6 mg/kg; Number of days free of MV; Test type: Superiority; p = 0.0130, One-sided p-value from re-randomization
Statistical Analysis 3: Comparison: Placebo vs recAP 1.6 mg/kg; Number of days free of RRT; Test type: Superiority; p = 0.0250, One-sided p-value from re-randomization
Statistical Analysis 4: Comparison: Placebo vs recAP 1.6 mg/kg; Number of days free of vasopressors and inotropes; Test type: Superiority; p = 0.0730, One-sided p-value from re-randomization

10. Secondary Outcome: Days Alive and Free of Organ Support Through Day 28: COVID-19 Population
Description: as for outcome 8
Time Frame: 28 days
Population: COVID-19 modified intent-to-treat Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | recAP 1.6 mg/kg
Number analyzed (Participants) | 13 | 20
days
  Days alive and free of organ support through to Day 28 | 1.5 (5.27) | 8.3 (10.24)
  Number of days free of MV | 3.3 (8.14) | 8.6 (10.85)
  Number of days free of RRT | 2.3 (7.74) | 19.7 (13.09)
  Number of days free of vasopressors and inotropes | 3.6 (8.83) | 14.9 (11.29)
Statistical Analysis 1: Comparison: Placebo vs recAP 1.6 mg/kg; Days alive and free of organ support through Day 28; Test type: Superiority; p = 1.0000, One-sided p-value from re-randomization
Statistical Analysis 2: Comparison: Placebo vs recAP 1.6 mg/kg; Number of days free of MV; Test type: Superiority; p = 0.9790, One-sided p-value from re-randomization
Statistical Analysis 3: Comparison: Placebo vs recAP 1.6 mg/kg; Number of days free of RRT; Test type: Superiority; p = 0.6750, One-sided p-value from re-randomization
Statistical Analysis 4: Comparison: Placebo vs recAP 1.6 mg/kg; Number of days free of vasopressors and inotropes; Test type: Superiority; p = 0.0310, One-sided p-value from re-randomization

11. Secondary Outcome: Days Alive and Out of the ICU Through Day 28: Main Trial Population
Description: Days alive and out of the ICU through Day 28 (with death within 28 days counting as zero days).
Time Frame: 28 days
Population: Main Trial modified intent-to-treat Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | recAP 1.6 mg/kg
Number analyzed (Participants) | 277 | 279
Days | 11.4 (10.56) | 11.4 (10.42)
Statistical Analysis 1: Comparison: Placebo vs recAP 1.6 mg/kg; Test type: Superiority; p = 0.5450, One-sided p-value from re-randomization

12. Secondary Outcome: Days Alive and Out of the ICU Through Day 28: Moderate Chronic Kidney Disease Population
Description: Days alive and out of the ICU through Day 28 (with death within 28 days counting as zero days).
Time Frame: 28 days
Population: Moderate Chronic Kidney Disease modified intent-to-treat Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | recAP 1.6 mg/kg
Number analyzed (Participants) | 31 | 30
Days | 8.1 (9.60) | 14.7 (10.09)
Statistical Analysis 1: Comparison: Placebo vs recAP 1.6 mg/kg; Test type: Superiority; p = 0.0810, One-sided p-value from re-randomization

13. Secondary Outcome: Days Alive and Out of the ICU Through Day 28: COVID-19 Population
Description: Days alive and out of the ICU through Day 28 (with death within 28 days counting as zero days).
Time Frame: 28 days
Population: COVID-19 modified intent-to-treat Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | recAP 1.6 mg/kg
Number analyzed (Participants) | 13 | 20
Days | 3.0 (7.39) | 7.5 (9.60)
Statistical Analysis 1: Comparison: Placebo vs recAP 1.6 mg/kg; Test type: Superiority; p = 0.9790, One-sided p-value from re-randomization

14. Secondary Outcome: 90-day All Cause Mortality: Main Trial Population
Description: 90-Day all-cause mortality
Time Frame: 90 days
Population: Main Trial modified intent-to-treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | recAP 1.6 mg/kg
Number analyzed (Participants) | 277 | 279
Participants
  Participants with event | 89 | 97
  Participants censored | 188 | 182
Statistical Analysis 1: Comparison: Placebo vs recAP 1.6 mg/kg; Test type: Superiority; p = 0.6916, One-sided p-value; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.806 to 1.437]

15. Secondary Outcome: 90-day All Cause Mortality: Moderate Chronic Kidney Disease Population
Description: 90-Day all-cause mortality
Time Frame: 90 days
Population: Moderate Chronic Kidney Disease modified intent-to-treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | recAP 1.6 mg/kg
Number analyzed (Participants) | 31 | 30
Participants
  Participants with event | 13 | 7
  Participants censored | 18 | 23
Statistical Analysis 1: Comparison: Placebo vs recAP 1.6 mg/kg; Test type: Superiority; p = 0.0628, One-sided p-value; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.180 to 1.234]

16. Secondary Outcome: 90-day All Cause Mortality: COVID-19 Population
Description: 90-Day all-cause mortality
Time Frame: 90 days
Population: COVID-19 modified intent-to-treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | recAP 1.6 mg/kg
Number analyzed (Participants) | 13 | 20
Participants
  Participants with event | 11 | 6
  Participants censored | 2 | 14
Statistical Analysis 1: Comparison: Placebo vs recAP 1.6 mg/kg; Test type: Superiority; p < 0.0001, One-sided p-value; Hazard Ratio (HR) = 0.01, 95% CI 2-sided [0.001 to 0.054]

ADVERSE EVENTS:
Time Frame: All AEs were followed to D28, inclusive. Ongoing SAEs on D28 were followed until resolution, deemed to be chronic or not clinically significant, or until the participant was considered stable or was lost to follow-up (up to D180). SAEs starting after D28 were to be reported if at least possibly related to study drug. Patients' mortality status was collected in a separate CRF module up to D180, or date of premature termination.
Description: In the safety population participants were analyzed according to treatment received.
Groups:
- Placebo (Main Trial Safety Population, n=276): Matching placebo; 3 daily 1-hour continuous intravenous infusions on Days 1, 2 and 3
  Main Trial Population: Participants with a pre-AKI reference eGFR greater than or equal to 45 mL/min/1.73 m2 and no proven or suspected COVID-19 at time of randomization
- recAP 1.6 mg/kg (Main Trial Safety Population, n=280): Recombinant human alkaline phosphatase (recAP) 1.6mg/kg; 3 daily 1-hour continuous intravenous infusions on Days 1, 2 and 3
  Main Trial Population: Participants with a pre-AKI reference eGFR greater than or equal to 45 mL/min/1.73 m2 and no proven or suspected COVID-19 at time of randomization
- Placebo (Moderate CKD Trial Safety Population, n=31): Matching placebo; 3 daily 1-hour continuous intravenous infusions on Days 1, 2 and 3.
  Moderate chronic kidney disease (CKD) Population: Participants with a pre-acute kidney injury reference estimated glomerular filtration rate more than or equal to 25 and less than 45 mL/min/1.73 m2 and no proven or suspected COVID-19 at time of randomization
- recAP 1.6 mg/kg (Moderate CKD Safety Population, n=30): Recombinant human alkaline phosphatase (recAP) 1.6mg/kg; 3 daily 1-hour continuous intravenous infusions on Days 1, 2 and 3 Moderate chronic kidney disease (CKD) Population: Participants with a pre-acute kidney injury reference estimated glomerular filtration rate more than or equal to 25 and less than 45 mL/min/1.73 m2 and no proven or suspected COVID-19 at time of randomization
- Placebo (Covid-19 Safety Population, n=13): Matching placebo; 3 daily 1-hour continuous intravenous infusions on Days 1, 2 and 3.
  COVID-19 Population: Participants with proven or suspected COVID-19 at time of randomization with or without 'moderate' chronic kidney disease and, for patients in this population, COVID-19 should have been the main cause of sepsis-associated acute kidney injury
- recAP 1.6 mg/kg (Covid-19 Safety Population, n=20): Recombinant human alkaline phosphatase (recAP) 1.6mg/kg; 3 daily 1-hour continuous intravenous infusions on Days 1, 2 and 3 COVID-19 Population: Participants with proven or suspected COVID-19 at time of randomization with or without 'moderate' chronic kidney disease and, for patients in this population, COVID-19 should have been the main cause of sepsis-associated acute kidney injury
Arm/Group | Placebo (Main Trial Safety Population, n=276) | recAP 1.6 mg/kg (Main Trial Safety Population, n=280) | Placebo (Moderate CKD Trial Safety Population, n=31) | recAP 1.6 mg/kg (Moderate CKD Safety Population, n=30) | Placebo (Covid-19 Safety Population, n=13) | recAP 1.6 mg/kg (Covid-19 Safety Population, n=20)
All-Cause Mortality (participants affected / at risk) | 92/276 | 108/280 | 14/31 | 7/30 | 11/13 | 7/20
Serious Adverse Events (participants affected / at risk) | 112/276 | 125/280 | 18/31 | 11/30 | 11/13 | 7/20
Other Adverse Events (participants affected / at risk) | 142/276 | 131/280 | 18/31 | 13/30 | 5/13 | 12/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Main Trial Safety Population, n=276) (N=276) | recAP 1.6 mg/kg (Main Trial Safety Population, n=280) (N=280) | Placebo (Moderate CKD Trial Safety Population, n=31) (N=31) | recAP 1.6 mg/kg (Moderate CKD Safety Population, n=30) (N=30) | Placebo (Covid-19 Safety Population, n=13) (N=13) | recAP 1.6 mg/kg (Covid-19 Safety Population, n=20) (N=20)
Septic shock (Infections and infestations) | 21 (21) | 16 (16) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 8 (10) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest wall abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex encephalitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Purulent pericarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungaemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 15 (15) | 0 (0) | 1 (1) | 5 (5) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 7 (8) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Torsade de pointes (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papillary muscle rupture (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 12 (12) | 16 (16) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Hernia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 4 (4) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mesenteric venous occlusion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Necrotising oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurological decompensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serotonin syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drain site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fascial rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear haemorrhage (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Schizoaffective disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mediastinal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspergillus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extradural abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus enterocolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Necrotising soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extremity necrosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatorenal failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Plasmablastic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intensive care unit acquired weakness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuromyopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Main Trial Safety Population, n=276) (N=276) | recAP 1.6 mg/kg (Main Trial Safety Population, n=280) (N=280) | Placebo (Moderate CKD Trial Safety Population, n=31) (N=31) | recAP 1.6 mg/kg (Moderate CKD Safety Population, n=30) (N=30) | Placebo (Covid-19 Safety Population, n=13) (N=13) | recAP 1.6 mg/kg (Covid-19 Safety Population, n=20) (N=20)
Hypokalaemia (Metabolism and nutrition disorders) | 12 (13) | 15 (15) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 9 (9) | 11 (11) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (4) | 8 (8) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (5) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 16 (17) | 26 (26) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 13 (14) | 12 (12) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 22 (23) | 26 (28) | 2 (3) | 3 (3) | 0 (0) | 3 (3)
Pneumonia (Infections and infestations) | 10 (11) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 10 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 5 (5) | 10 (10) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 12 (13) | 8 (10) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 7 (7) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 11 (12) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 3 (3) | 4 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (4) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 2 (2) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 2 (2) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Penile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal wall infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea cruris (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ulcerative gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemodynamic instability (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intensive care unit acquired weakness (Nervous system disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileostomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toe amputation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood lactic acid increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric residual increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterococcus test positive (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial was terminated early due to futility being reached for the primary endpoint of all cause mortality at day 28 at the interim analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/72/NCT04411472/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/72/NCT04411472/SAP_001.pdf